CLINICAL TRIAL: NCT02776410
Title: Young Consumers' Attitudes and Behaviour Towards Sustainable and Healthy Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zuzanna Pieniak (Other)
Collaborators: National Science Centre, Poland (Other Government)
Responsible Party: Sponsor-Investigator, Zuzanna Pieniak, phd, Consumer and Sensory Research Institute Ltd, Poland
Organization: Consumer and Sensory Research Institute Ltd, Poland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2013/10/M/HS4/00477
Record Dates: First submitted 2016-05-12; First posted 2016-05-18 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Sustainable Healthy Eating Behaviour
Keywords: sustainable healthy eating; consumer behaviour; consumer attitudes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Group receiving tailored messages promoting sustainable and healthy eating through an mobile-application together with six principles of sustainable healthy eating that will be included in the mobile application,
  Interventions: Behavioral: Consumer reactions to tailored messages sent via app
- Control group (No Intervention): Group who will not download the mobile application

INTERVENTIONS:
Behavioral: Consumer reactions to tailored messages sent via app — The intervention will take 1 month. Participants from the Intervention group will receive tailored messages every 2-3 days with a push notification. Additionally, interaction with the participants via the use of app is foreseen.
  Arms: Intervention group

SUMMARY:
The purpose is to investigate young consumers' attitudes and behaviour towards sustainable and healthy eating by applying a multidisciplinary approach, taking into account economical, marketing, public health and environmental related issues. In order to achieve this goal, consumers' reactions on interactive tailored informational messages about sustainable from social, environmental and economical point of view, as well as healthy eating behaviour in a group of Polish young adults will be investigated. Main research questions that will be addressed: What is consumer's current behaviour and perception of sustainable healthy eating? What are factors determining consumers' reactions to messages about sustainable healthy eating? What are consumers' reactions on interactive tailored communication about sustainable and healthy eating behaviour? About 200 Polish consumers will take part in this randomized controlled trial. A stratified design will be used to recruit 18-30 years old adults using smart phones. The sample will be represented for gender and region. Participants will be randomly assigned to either a study or a control group. They will complete a baseline and follow-up survey. An application for smart phones will be developed by a professional IT company in order to deliver personalised messages to the participants. Intervention will take one month. Messages developed following the theory-linked definitions of behaviour change techniques will be sent to the participants every 2-3 days. The six principles of sustainable and healthy behaviour introduced in the campaign "Livewell 2020" will be used as a base to communicate to consumers.

ELIGIBILITY:
Inclusion Criteria:

* user of a smart phone
* Internet user

Exclusion Criteria:

* user of an older version of a mobile phone

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 201 (Actual)
Dates: Start 2016-05; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
change in sustainable healthy eating behaviour measured by a Sustainable Healthy Eating index | baseline and follow up 2 months later

SECONDARY OUTCOMES:
consumer attitudes towards sustainable healthy eating | baseline and follow up 2 months later
  consumer attitudes towards sustainable healthy eating by means of quantitative questionnaire at the baseline survey prior to intervention and follow up survey after the intervention
consumer knowledge about sustainable healthy eating | baseline and follow up 2 months later
  consumer subjective and objective knowledge about sustainable healthy eating by means of scales as a part of the quantitative questionnaire at the baseline survey prior to intervention and follow up survey after the intervention
Intention towards sustainable healthy eating | baseline and follow up 2 months later
  Intention towards sustainable healthy eating by means of a scale as a part of the quantitative questionnaire at the baseline survey prior to intervention and follow up survey after the intervention
Behavioural determinants of sustainable healthy eating based on the Integrative Model | baseline and follow up 2 months later
  Other behavioural determinants of sustainable healthy eating by means of quantitative questionnaire at the baseline survey prior to intervention and follow up survey after the intervention

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pieniak Z, Zakowska-Biemans S, Kostyra E, Raats M. Sustainable healthy eating behaviour of young adults: towards a novel methodological approach. BMC Public Health. 2016 Jul 15;16:577. doi: 10.1186/s12889-016-3260-1. PMID 27421759